CLINICAL TRIAL: NCT07240662
Title: Vorasidenib in CNS WHO Grade 2 IDH-mutant Diffuse Glioma: A Multicenter, Prospective, Non-interventional Study in Germany
Brief Title: Vorasidenib in CNS WHO Grade 2 IDH-mutant Diffuse Glioma
Acronym: VIOLETA
Status: Recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-120529
Record Dates: First submitted 2025-09-29; First posted 2025-11-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Glioma
Keywords: WHO Grade 2; IDH-mutant; diffuse
MeSH Terms: conditions — Glioma | interventions — vorasidenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Vorasidenib — oral, first-in-class, dual inhibitor of mIDH 1 and 2

SUMMARY:
The goal of this prospective, observational study VIOLETA is to collect real-world data on vorasidenib treatment in a broad patient population. Though vorasidenib can be administered from 12 years old, VIOLETA focuses on adult patients with IDH1- or IDH2-mutant WHO grade 2 glioma who receive vorasidenib following surgery according to the current SmPC. Thus, VIOLETA will evaluate for the first-time treatment with vorasidenib in German clinical routine. To gain knowledge about how vorasidenib treatment affects patients' well-being, the primary objective of the study is to assess patients' quality of life. Further patient-relevant endpoints addressed by this study will include seizure burden, PFS, Objective Response Rate (ORR), TTNI, safety as well as factors affecting treatment decision making.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* WHO grade 2 astrocytoma or oligodendroglioma
* Presence of IDH1- or IDH2-mutation
* Surgical intervention
* No immediate need of radiotherapy or chemotherapy according to the treating physician
* Decision for treatment with vorasidenib as per current SmPC
* Signed written informed consent*
* Willingness to participate in Patient-Reported Outcome (PRO) assessment in German language
* Other criteria according to current SmPC * Patients are allowed to be enrolled up to 6 weeks after their first intake of vorasidenib but must still be on treatment at the time of enrollment

Exclusion Criteria:

* Participation in an interventional clinical trial
* Patient unable to consent
* Other contraindications according to current SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (at least 40 kg) with predominantly non-enhancing grade 2 astrocytoma or oligodendroglioma with an IDH1 or IDH2 mutation who only had surgical intervention and are not in immediate need of radiotherapy or chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate Quality of Life (QoL) by the Functional Assessment of Cancer Therapy - Brain (FACT-Br) questionnaire over the course of treatment | baseline, up to 72 months
  Evaluate QoL by the FACT-Br questionnaire over the course of treatment. Change from baseline in the FACT-Br total score over time. The FACT-Br total score ranges from 0 to 200, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Evaluate Quality of Life (QoL) by using the Functional Assessment of Cancer Therapy - Brain (FACT-Br) questionnaire at start and during course of vorasidenib treatment | baseline, up to 72 months
  Evaluate QoL by using the FACT-Br questionnaire at start and during course of vorasidenib treatment. Change from baseline over time for all other scales of the FACT-Br. For all scales, the higher the score the better quality of life.
Assess seizure activity and severity at baseline and during treatment: Proportion of patients with baseline seizure activity | baseline, up to 72 months
  Proportion of patients with baseline seizure activity is defined as at least 1 seizure in the previous 30 days prior to vorasidenib treatment start
Assess seizure activity and severity at baseline and during treatment: event rate of seizures | baseline, up to 72 months
  Exposure adjusted event rate of seizures according to patient-reported outcome (patient diary)
Assess seizure activity and severity at baseline and during treatment: event rate of seizures with loss of consciousness | baseline, up to 72 months
  Exposure adjusted event rate of seizures with loss of consciousness according to PRO (patient diary)
Assess seizure activity and severity at baseline and during treatment: incidence rate of seizures | baseline, up to 72 months
  Exposure adjusted incidence rate of seizures according to patient-recorded outcome
Assess seizure activity and severity at baseline and during treatment: incidence rate of seizures with loss of consciousness | baseline, up to 72 months
  Exposure adjusted incidence rate of seizures according to patient-reported outcome
Assess seizure activity and severity at baseline and during treatment: Change from baseline of seizures | max. 72 months; from patient-specific study start to end of study (during vorasidenib treatment and follow-up)
  Change from baseline of seizures reported by the patients during course of treatment
Assess seizure activity and severity at baseline and during treatment: Change from baseline of seizures with loss of consciousness | baseline, up to 72 months
  Change from baseline of seizures with loss of consciousness reported by the patients during course of treatment
Assess effectiveness in routine treatment: Progression-free survival | baseline, up to 72 months
  PFS ist defined as time interval measured from the day of first vorasidenib administration to first progression or death, whichever comes first. Patients without tumor progression or death at the time of analysis will be censored at their date of last contact.
Assess effectiveness in routine treatment: Overall Survival (OS) | baseline, up to 72 months
  OS is defined as the time interval measured form the day of first vorasidenib administration to time of death from any cause. Time to last contact will be used if a patient has no documented date of death and OS for the patient will be considered censored.
Assess effectiveness in routine treatment: Objective response rate (ORR) | max. 72 months; from patient-specific study start to end of study (during vorasidenib treatment and follow-up)
  ORR is defined as the proportion of patients achieving Complete Response (CR), Partial Response (PR), or Minor Response (MR) as best response.
Assess effectiveness in routine treatment: Disease Control Rate (DCR) | baseline, up to 72 months
  DCR is defined as proportion of patients with Complete Response, Partial Response, Minor Response or Stable Disease as best response.
Assess effectiveness in routine treatment: Best response | baseline, up to 72 months
  Best response is defined as Complete Response (CR), Partial Response (PR), Minor Response (MR), Stable Disease (SD), or Progressive Disease (PD))
Assess effectiveness in routine treatment: Time to next intervention (TTNI) | baseline, up to 72 months
  Time to next intervention is defined as time from first administration of vorasidenib until initiation of next intervention (i.e., subsequent antineoplastic treatment, surgery, chemotherapy or radiotherapy) or death, whichever comes first.
Assess drug safety: Incidence of (serious) adverse events ((S)AEs) | Baseline up to 30 days after vorasidenib treatment
  Incidence of (serious) AEs ((S)AEs) as characterized by type, frequency, severity and seriousness.
Assess drug safety: Incidence of (serious) adverse drug reactions ((S)ADRs) | Baseline up to 30 days after vorasidenib treatment
  Incidence of (serious) adverse drug reactions ((S)ADRs) as characterized by type, frequency, severity and seriousness.
Assess drug safety: Incidence of seizures reported as treatment-emergent adverse events (TEAEs) | Baseline up to 30 days after vorasidenib treatment
  Treatment-emergent adverse events (TEAE) are adverse events that were not present before medical treatment, or a pre-existing event that worsens in intensity or frequency during vorasidenib treatment and the following 30 days.
Assess parameters of physicians' treatment decision making using a questionnaire | Baseline
  Frequency of distinct parameters affecting therapy choice; questionnaire completed by treating physician.
Duration of treatment with vorasidenib | baseline, up to 72 months
  Describe treatment reality in detail: Duration of treatment with vorasidenib
Frequency of treatment modifications with reasons | baseline, up to 72 months
  Describe treatment reality in detail: Frequency of treatment modifications with reasons
Time to start of vorasidenib treatment after initial diagnosis | Baseline
  Describe treatment reality in detail: Time to start of vorasidenib treatment after initial diagnosis
Time to start of vorasidenib treatment after surgery | Baseline
  Describe treatment reality in detail: Time to start of vorasidenib treatment after surgery
Frequency of distinct subsequent antineoplastic therapies (systemic therapies including substances, surgeries, radiotherapies) | baseline, up to 72 months
  Describe treatment reality in detail: Frequency of distinct subsequent antineoplastic therapies (systemic therapies including substances, surgeries, radiotherapies)
Anti-epileptic medication: Proportion of patients with anti-epileptic drug (AED) treatment at baseline | baseline, up to 72 months
  Proportion of patients with anti-epileptic drug treatment at baseline (i.e. 30 days prior treatment)
Anti-epileptic medication: Proportion of patients with AED treatment during treatment | baseline, up to 72 months
  Proportion of patients with anti-epileptic drug treatment during treatment
Anti-epileptic medication: Type of AED | baseline, up to 72 months
  Anti-epileptic medication during course of treatment
Anti-epileptic medication: Doses of AED | baseline, up to 72 months
  Doses of anti-epileptic medication over the course of time
Anti-epileptic medication: AED modifications | baseline, up to 72 months
  Type of anti-epileptic medication modifications
Anti-epileptic medication: Reasons for AED modifications | baseline, up to 72 months
  Anti-epileptic medication modifications with reasons thereof
Anti-epileptic medication: Frequency of patients under AED treatment after End of Treatment (EOT) of vorasidenib | from end of treatment to end of study, up to 72 months
  Frequency of patients under AED treatment after EOT of vorasidenib (incl. dose)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationales Centrum für Tumorerkrankungen (NCT) Heidelberg, Heidelberg, Germany